CLINICAL TRIAL: NCT02601794
Title: Delivering an Intervention to Accompany Supportive Care
Brief Title: A Study of Delivering a Mindfulness App Intervention to Accompany Supportive Care Among Women With Breast Cancer
Acronym: DIVAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Suyen Warzinski, Research Scientist, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC20140010H
Record Dates: First submitted 2015-11-04; First posted 2015-11-10 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; mHealth; Mindfulness; Complementary Therapies
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- App-based Mindfulness Training (Experimental): 12 week mindfulness training delivered remotely through mobile app
  Interventions: Behavioral: App-based Mindfulness Training
- Waitlist Control (No Intervention): No intervention provided during study period. 12 week mindfulness training will be delivered through mobile app once all study assessments have been completed

INTERVENTIONS:
Behavioral: App-based Mindfulness Training — A commercially available mindfulness training app delivered to smartphone or tablet.
  Other Names: AMT
  Arms: App-based Mindfulness Training

SUMMARY:
The investigators are conducting a web-based study to explore the use of a mindfulness app to improve quality of life among women with breast cancer.

Eligible participants will be asked to provide informed consent to participate and submit a data authorization form to obtain information from the app at the end of the project.

This 12-week project will randomly assign participants to one of two groups:

Group 1 (AMT) will receive the mindfulness app right away; Group 2 (WC) will receive the mindfulness app at the end of 12 weeks.

All participants will receive a welcome email with group designation. Participants assigned to Group 1 (AMT) will also receive app download instructions and pass code. Group 1 will be asked to complete the app's first 10-minute mindfulness exercise, at minimum.

Participants assigned to Group 2 (WC) will be notified that they will receive app download instructions and pass code at the end of 12 weeks.

Regardless of group assignment, all participants will be asked to complete web-based survey assessments 4 different times throughout the study (baseline, week 5, week 9, 12-week follow up). The surveys will be related to quality of life, mindfulness, mobile technology, health literacy, and chronic pain.

To encourage participation, a member of the study team will send out weekly check-in emails.

Once all data has been collected, app developers will provide the investigators with app data for each participant, including times accessed, length of time using app. This information will help the investigators observe which app characteristics are most useful, as well as the optimal amount of time needed to obtain benefit from the app.

The investigators goals are to understand how using the mindfulness app compares to not using the mindfulness app. The investigators will also observe whether the app contributes to participants' quality of life. The investigators also want to understand more about how women use health apps overall. This information may inform issues related to delivery of app-based health interventions among women with breast cancer.

DETAILED DESCRIPTION:
The proposed project utilizes a randomized controlled trial design to explore the efficacy of a commercial app-based mindfulness training (AMT) intervention for women with breast cancer, compared to waitlist control (WC).

Recruitment commenced in August 2015 and will continue until March 2016. Up to 180 participants will be recruited using a combination recruitment strategy, including social media, word of mouth, registries, and informing colleagues of the project. The proposed sample size, powered to detect changes in quality of life, is adequate for 70% power, while accounting for attrition.

Eligible participants will be randomly assigned to app-based mindfulness training (AMT; n=90) or waitlist control (WC; n=90). Group assignment will be stratified by endorsement of past year mind-body complementary or alternative medicine practice indicated at baseline.

Informed consent will be obtained at baseline, prior to completion of assessments. Participants will also be asked to sign a data authorization allowing the research team to obtain app metadata at the completion of the study:

At baseline (pre-group assignment), participants will be required to complete web-based survey assessments related to quality of life, mindfulness, health literacy, health apps, and chronic pain. A unique web link to a secure data collection website will be emailed to each participant. Participants will have up to 7 days to complete assessments. Group assignment will be ongoing, as participants enroll.

All participants completing baseline assessments will receive a welcome email indicating group assignment. Participants assigned to AMT will receive app download instructions and pass code in the welcome email.

All participants will receive weekly check-in emails to facilitate engagement and retention.

At week 5 and week 9, all participants will complete web-based survey assessments related to quality of life, mindfulness, and chronic pain. A fidelity check will be completed to identify group contamination or new use of other health apps.

At 12-week follow up, all participants will complete web-based survey assessments related to quality of life, mindfulness, and chronic pain. A fidelity check will be completed to identify group contamination or new use of other health apps. At this time, participants assigned to WC will receive app download instructions and pass code.

At the study completion, app developers will provide the investigators with app log data at the individual level. This information will help the investigators observe which app characteristics are most useful, as well as the optimal amount of time needed to obtain benefit from the app.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age ≥ 25
3. Breast cancer diagnosis within past 5 years
4. Willing to provide locator information for follow-up contact
5. Reliable internet access
6. Ownership of smartphone or tablet with following specifications: wireless capability, running on iOS or Android operating system, current software (4.4 Android; 8.0 iOS or later), and adequate memory to run the mindfulness app (43M Android; 30.2M iOS).

Exclusion Criteria:

1. Unfamiliar with mobile phones/tablets, including ability to download and register mindfulness app
2. Become unable to participate in a fully app and web-based intervention trial
3. Unwilling to complete online questionnaires
4. Unwilling to use personal phone/tablet to test intervention

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in breast cancer-related quality of life scores | Change from baseline FACT-B scores at 12 weeks
  Measured by the Functional Assessment of Cancer Therapy-Breast (FACT-B)

SECONDARY OUTCOMES:
Change in mindfulness scores | Change from baseline MAAS scores at 12 weeks
  Measured by the Mindful Attention Awareness Scale (MAAS)
Change in spiritual quality of life scores | Change from baseline FACIT-SP scores at 12 weeks
  Measured by the Functional Assessment of Chronic Illness Therapy (FACIT-SP)

OTHER OUTCOMES:
Change in pain-related severity and interference | Change from baseline BPI scores at 12 weeks
  Measured by the Brief Pain Inventory (BPI)
App usability | Measured at 5 weeks
  Measured by the Systems Usability Scale
eHealth literacy scores | Measured at baseline
  Measured by the eHealth Literacy Scale (eHEALS)
Health literacy scores | Measured at baseline
  Measured by the Brief Health Literacy Screen

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Rosen, MPH, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- University of Texas Health Science Center San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Peterman AH, Fitchett G, Brady MJ, Hernandez L, Cella D. Measuring spiritual well-being in people with cancer: the functional assessment of chronic illness therapy--Spiritual Well-being Scale (FACIT-Sp). Ann Behav Med. 2002 Winter;24(1):49-58. doi: 10.1207/S15324796ABM2401_06. PMID 12008794
- [Background] Brooke J. SUS: a "quick and dirty" usability scale. In Jordan PW, Thomas B, McClelland IL, Weerdmeester B, eds. Usability Evaluation In Industry. Boca Raton: CRC Press; 1996:189-94.
- [Background] Brady MJ, Cella DF, Mo F, Bonomi AE, Tulsky DS, Lloyd SR, Deasy S, Cobleigh M, Shiomoto G. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. J Clin Oncol. 1997 Mar;15(3):974-86. doi: 10.1200/JCO.1997.15.3.974. PMID 9060536
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Norman CD, Skinner HA. eHEALS: The eHealth Literacy Scale. J Med Internet Res. 2006 Nov 14;8(4):e27. doi: 10.2196/jmir.8.4.e27. PMID 17213046
- [Background] Haun J, Noland-Dodd V, Varnes J, Graham-Pole J, Rienzo B, Donaldson P. Testing the BRIEF health literacy screening tool. Federal Practitioner 26(12): 24-31, 2009.